CLINICAL TRIAL: NCT02782806
Title: Spot-Check Noninvasive Hemoglobin (SpHb) Clinical Validation
Brief Title: Spot-Check Noninvasive Pulse CO-Oximeter Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TORR0001
Record Dates: First submitted 2016-05-12; First posted 2016-05-25 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Anemia
Keywords: Noninvasive; Pulse; CO-Oximeter; Validation
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes

ARMS (1):
- Test group (Experimental): All subjects are enrolled into the test group and receive Masimo Rad-67 Pulse Oximeter for measurement of hemoglobin.
  Interventions: Device: Masimo Rad-67 Pulse Oximeter

INTERVENTIONS:
Device: Masimo Rad-67 Pulse Oximeter — Noninvasive pulse oximeter

SUMMARY:
In this study, the accuracy of a noninvasive hemoglobin sensor(s) will be assessed by comparison to hemoglobin measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: Greater than one month
* Weight: Greater than or equal to 3kg
* Any racial or ethnic group
* The subject or the subject's legally authorized representative has given written informed consent/assent to participate in the study
* If an ICU patient, total hemoglobin of < 9 g/dL at time of screening.

Exclusion Criteria:

* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as burns, scar tissue, nail polish, acrylic nails, infections, abnormalities, etc.
* Subjects deemed not suitable for the study at the discretion of the investigator
* Subjects unlikely to be able to refrain from excessive motion during data collection. Excessive motion includes postural changes, making hand gestures, involuntary muscular movements, etc.

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Accuracy of sensor | Up to 1 hr per subject
  Accuracy willl be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States